CLINICAL TRIAL: NCT02105688
Title: A Phase III Randomized Clinical Trial to Study the Efficacy and Safety of the Combination Regimen of MK-5172/MK-8742 in Treatment-Naïve Subjects With Chronic HCV GT1, GT4, and GT6 Infection Who Are on Opiate Substitution Therapy
Brief Title: An Efficacy and Safety Study of Grazoprevir (MK-5172) + Elbasvir (MK-8742) in the Treatment of Chronic Hepatitis C Virus (HCV) Genotype (GT)1, 4, or 6 Infection in Treatment-Naïve Participants Who Are on Opiate Substitution Therapy (MK-5172-062)
Acronym: C-EDGE CO-STAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5172-062; 2014-000343-32 (EudraCT Number); MK-5172-062 (Other: Merck)
Record Dates: First submitted 2014-04-02; First posted 2014-04-07 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2019-11

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — grazoprevir; elbasvir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Treatment Arm: Grazoprevir/Elbasvir (Experimental): In Part A, participants receive grazoprevir 100 mg plus elbasvir 50 mg FDC (MK-5172A) once daily for 12 weeks (blinded) and were followed-up for 24 weeks. In Part B, participants could enroll in a 3-year follow-up period where they were followed every 6 months for 3 years in an observational cohort (no treatment was administered during Part B).
  Interventions: Drug: Grazoprevir 100 mg/Elbasvir 50 mg FDC tablet (MK-5172A)
- Deferred Treatment Arm: Placebo > Grazoprevir/Elbasvir (Placebo Comparator): In Part A, participants receive placebo to MK-5172A once daily for 12 weeks (blinded), followed by 4 weeks of follow-up. Afterwards, participants received 12 weeks of open-label treatment with the MK-5172A FDC and were followed-up for 24 weeks. In Part B, participants could enroll in a 3-year follow-up period where they were followed every 6 months for 3 years in an observational cohort (no treatment was administered during Part B).
  Interventions: Drug: Grazoprevir 100 mg/Elbasvir 50 mg FDC tablet (MK-5172A); Drug: Placebo to Grazoprevir 100 mg/Elbasvir 50 mg FDC tablet

INTERVENTIONS:
Drug: Grazoprevir 100 mg/Elbasvir 50 mg FDC tablet (MK-5172A) — Grazoprevir 100 mg/Elbasvir 50 mg FDC tablet, taken once daily by mouth for 12 weeks.
  Other Names: MK-5172A
Drug: Placebo to Grazoprevir 100 mg/Elbasvir 50 mg FDC tablet — Placebo Grazoprevir 100 mg/Elbasvir 50 mg FDC tablet, taken once daily by mouth for 12 weeks.
  Arms: Deferred Treatment Arm: Placebo > Grazoprevir/Elbasvir

SUMMARY:
This is a 2-part study. The purpose of Part A is to assess the efficacy and safety of grazoprevir (MK-5172) 100 mg in combination with elbasvir (MK-8742) 50 mg for 12 weeks in the treatment of chronic HCV GT1, GT4, or GT6 infection in treatment-naïve participants who are on opiate substitution therapy (OST). The primary hypothesis is that the percentage of participants who receive grazoprevir/elbasvir fixed-dose combination (FDC) in the Immediate Treatment Arm and achieve a Sustained Virologic Response 12 weeks after the end of all study therapy (SVR12) will be superior to 67%. In addition, participants who received at least 1 dose of grazoprevir/elbasvir in Part A will be eligible to participate in Part B, which is a 3-year observational follow-up.

ELIGIBILITY:
Inclusion Criteria:

Part A

* Documented chronic HCV GT1, GT4, or GT6 infection with no evidence of GT2, GT3, GT5 or non-typeable genotypes and HCV ribonucleic acid (RNA) confirmed by screening lab results prior to randomization
* On opiate substitution therapy (OST; methadone, levamethadone, buprenorphine, naloxone, naltrexone) for at least 3 months prior to screening
* Treatment naïve to all HCV therapies
* Human Immunodeficiency Virus (HIV)-infected participants enrolled in this study must meet following criteria:
* Documented HIV infection
* Naïve to treatment with any antiretroviral therapy (ART) OR on HIV ART for at least 8 weeks prior to study entry using a dual nucleoside reverse transcriptase inhibitor (NRTI) backbone of tenofovir or abacavir and either emtricitabine or lamivudine PLUS raltegravir (or dolutegravir or rilpivirine). Dose modifications or changes in ART during the 4 weeks prior to study entry (Day 1) are not permitted
* Cluster of differentiation 4 (CD4+) T-cell count >200 cells/mm^3 if on ART or >500 cell/mm^3 if ART treatment naïve
* Undetectable plasma HIV-1 RNA at least 8 weeks prior to screening if on ART or <50,000 copies/mL if ART treatment naïve
* Participants with HIV-1 infection and on ART must have at least one viable antiretroviral regimen alternative beyond their current regimen in the event of HIV virologic failure or the development of anti-retroviral drug resistance
* Females who are of reproductive potential must agree to avoid becoming pregnant while receiving study drug and for 14 days after the last dose of study drug by complying with one of the following: (1) practice abstinence from heterosexual activity OR (2) use (or have her partner use) acceptable contraception during heterosexual activity

Part B

* Received at least one dose of grazoprevir in combination with elbasvir in Part A. Receiving OST and keeping >80% of scheduled appointments while on OST were not required for Part B.

Exclusion Criteria:

Part A

* Evidence of decompensated liver disease
* For participants with cirrhosis, participants who are Child-Pugh Class B or C or who have a Pugh-Turcotte (CPT) score >6
* Is co-infected with hepatitis B virus
* Has cirrhosis and liver imaging within 6 months of Day 1 showing evidence of hepatocellular carcinoma (HCC) or is under evaluation for HCC
* Currently using or intends to use barbiturates during the treatment period of this study
* Is a female and is pregnant or breast-feeding, or expecting to conceive or donate eggs from Day 1 or anytime during treatment, and 14 days after the last dose of study medication, or longer if dictated by local regulations
* Any medical condition requiring or likely to require chronic systemic administration of corticosteroids, Tumor Necrosis Factor (TNF) antagonists, or other immunosuppressant drugs during the course of the trial
* Evidence or history of chronic hepatitis not caused by HCV

Part B

* Mentally or legally incapacitated, has significant emotional problems at the time of pre-study screening visit or expected during the conduct of the study or has a history of a clinically significant psychiatric disorder which, in the opinion of the investigator, would interfere with the study procedures
* Has a medical condition or personal circumstance which, in the opinion of the investigator and/or Sponsor, places the participant at unnecessary risk through continued participation in the trial or does not allow the participant to adhere to the requirements of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2014-09-02 (Actual); Primary Completion 2015-06-10 (Actual); Study Completion 2018-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Dore GJ, Altice F, Litwin AH, Dalgard O, Gane EJ, Shibolet O, Luetkemeyer A, Nahass R, Peng CY, Conway B, Grebely J, Howe AY, Gendrano IN, Chen E, Huang HC, Dutko FJ, Nickle DC, Nguyen BY, Wahl J, Barr E, Robertson MN, Platt HL; C-EDGE CO-STAR Study Group. Elbasvir-Grazoprevir to Treat Hepatitis C Virus Infection in Persons Receiving Opioid Agonist Therapy: A Randomized Trial. Ann Intern Med. 2016 Nov 1;165(9):625-634. doi: 10.7326/M16-0816. Epub 2016 Aug 9. PMID 27537841
- [Derived] Grebely J, Dore GJ, Altice FL, Conway B, Litwin AH, Norton BL, Dalgard O, Gane EJ, Shibolet O, Nahass R, Luetkemeyer AF, Peng CY, Iser D, Gendrano IN, Kelly MM, Hwang P, Asante-Appiah E, Haber BA, Barr E, Robertson MN, Platt H. Reinfection and Risk Behaviors After Treatment of Hepatitis C Virus Infection in Persons Receiving Opioid Agonist Therapy : A Cohort Study. Ann Intern Med. 2022 Sep;175(9):1221-1229. doi: 10.7326/M21-4119. Epub 2022 Aug 9. PMID 35939812
- [Derived] Asselah T, Reesink H, Gerstoft J, de Ledinghen V, Pockros PJ, Robertson M, Hwang P, Asante-Appiah E, Wahl J, Nguyen BY, Barr E, Talwani R, Serfaty L. Efficacy of elbasvir and grazoprevir in participants with hepatitis C virus genotype 4 infection: A pooled analysis. Liver Int. 2018 Sep;38(9):1583-1591. doi: 10.1111/liv.13727. Epub 2018 Mar 31. PMID 29461687
- [Derived] Reau N, Robertson MN, Feng HP, Caro L, Yeh WW, Nguyen BT, Wahl J, Barr E, Hwang P, Klopfer SO. Concomitant proton pump inhibitor use does not reduce the efficacy of elbasvir/grazoprevir: A pooled analysis of 1,322 patients with hepatitis C infection. Hepatol Commun. 2017 Aug 22;1(8):757-764. doi: 10.1002/hep4.1081. eCollection 2017 Oct. PMID 29404492

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 301 participants were randomized to either the Immediate Treatment Arm or to the Deferred Treatment Arm during Part A. 199 participants who completed Part A were enrolled in Part B; of these, 142 participants completed the study.
Groups:
- Immediate Treatment Arm: Grazoprevir/Elbasvir: In Part A, participants received grazoprevir 100 mg plus elbasvir 50 mg FDC (MK-5172A) once daily for 12 weeks (blinded) and were followed-up for 24 weeks. In Part B, participants could enroll in a 3-year follow-up period where they were followed every 6 months for 3 years in an observational cohort (no treatment was administered during Part B).
- Deferred Treatment Arm: Placebo > Grazoprevir/Elbasvir: In Part A, participants received placebo to MK-5172A once daily for 12 weeks (blinded), followed by 4 weeks of follow-up. Afterwards, participants received 12 weeks of open-label treatment with the MK-5172A FDC and were followed-up for 24 weeks. In Part B, participants could enroll in a 3-year follow-up period where they were followed every 6 months for 3 years in an observational cohort (no treatment was administered during Part B).
Period: Part A: Double-Blind
Arm/Group | Immediate Treatment Arm: Grazoprevir/Elbasvir | Deferred Treatment Arm: Placebo > Grazoprevir/Elbasvir
Started | 201 | 100
Completed | 181 (Completed Part A) | 83 (Completed Part A)
Not Completed | 20 | 17
Not completed — Adverse Event | 1 | 0
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 15 | 11
Not completed — Physician Decision | 0 | 1
Not completed — Status Unknown | 0 | 2
Not completed — Withdrawal by Subject | 4 | 2
Period: Part B: Observational Follow-up
Arm/Group | Immediate Treatment Arm: Grazoprevir/Elbasvir | Deferred Treatment Arm: Placebo > Grazoprevir/Elbasvir
Started | 131 (Completed Part A and met Part B Extension criteria) | 68 (Completed Part A and met Part B Extension criteria)
Completed | 94 (Completed Part B extension) | 48 (Completed Part B extension)
Not Completed | 37 | 20
Not completed — Death | 2 | 1
Not completed — Lost to Follow-up | 23 | 15
Not completed — Withdrawal by Subject | 9 | 3
Not completed — Physician Decision | 3 | 1

BASELINE CHARACTERISTICS:
Population: Baseline (BL) characteristics were reported for the Full Analysis Set (FAS): all randomized participants receiving ≥1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Treatment Arm: Grazoprevir/Elbasvir | Deferred Treatment Arm: Placebo > Grazoprevir/Elbasvir | Total
Number analyzed (Participants) | 201 | 100 | 301
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (9.9) | 46.4 (9.9) | 47.1 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 23 | 71
  Male | 153 | 77 | 230

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virologic Response 12 Weeks After the End of All Study Therapy (SVR12)
Description: Blood was drawn from each participant to assess Hepatitis C Virus ribonucleic acid (HCV RNA) plasma levels using the Roche COBAS® AmpliPrep/COBAS® Taqman HCV Test, v2.0, which had a lower limit of quantification of 15 IU/mL. SVR12 was defined as HCV RNA below the lower limit of detection (<LLOQ) at 12 weeks after the end of all study therapy for baseline infection, or HCV RNA≥ LLOQ demonstrated to be due to reinfection (after clearance of baseline infection). The Clopper-Pearson method was used to construct 95% confidence intervals for the SVR12 rate. The primary efficacy analysis for Part A was the percentage of participants in the immediate treatment arm (ITA) who achieved SVR12. SVR12 was also calculated for the Deferred Treatment Arm.
Time Frame: 12 weeks after end of all therapy (Study Week 24 for Immediate Treatment Arm and Study Week 40 for Deferred Treatment Arm)
Population: Modified FAS (mFAS): All randomized participants receiving ≥1 dose of active study treatment and excluding participants for study discontinuation for reasons unrelated to treatment regimen, response to HCV treatment, or BL genotype (GT)2, GT3, or GT5. The primary efficacy hypothesis was evaluated within participants of the Immediate Treatment Arm.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Immediate Treatment Arm: Grazoprevir/Elbasvir | Deferred Treatment Arm: Placebo > Grazoprevir/Elbasvir
Number analyzed (Participants) | 198 | 88
Percentage of Participants | 95.5 [91.5 to 97.9] | 96.6 [90.4 to 99.3]
Statistical Analysis 1: Comparison: Immediate Treatment Arm: Grazoprevir/Elbasvir; A one-sided exact test was used to test the null hypothesis, which was that the SVR12 rate for the ITA was less than 67% (historical reference rate derived from NCT01667731). The p-value was based on a one-sided exact test for a binomial proportion. A one-sided p-value <0.025 supports a conclusion that the true SVR12 is >67%; Test type: Superiority or Other; p < 0.001, One-sided exact test

2. Primary Outcome: Percentage of Participants Experiencing at Least One Adverse Event (AE) During the Double-Blind (DB) Treatment Period and First 14 Follow-up Days
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product, was also an AE. For this outcome measure, the primary safety analysis compared the percentage of participants experiencing an AE in the Immediate Treatment Arm during the double-blinded active treatment period to that of the Deferred Treatment Arm during the double-blinded placebo treatment period.
Time Frame: DB Treatment period plus first 14 follow-up days (up to Study Week 14)
Population: All randomized participants who received at least one dose of study treatment during the Part A DB period.
Measure: Number; unit: Percentage of Participants
Arm/Group | Immediate Treatment Arm: Grazoprevir/Elbasvir | Deferred Treatment Arm: Placebo > Grazoprevir/Elbasvir
Number analyzed (Participants) | 201 | 100
Percentage of Participants | 83.1 | 83.0
Statistical Analysis 1: Comparison: Immediate Treatment Arm: Grazoprevir/Elbasvir vs Deferred Treatment Arm: Placebo > Grazoprevir/Elbasvir; Categorical AE parameters were assessed via point estimates with 95% confidence intervals provided for between-treatment differences in the percentage of participants with events using the Miettinen and Nurminen method, an unconditional, asymptotic method; Test type: Superiority or Other; Difference in Percentage = 0.2, 95% CI 2-sided [-8.3 to 10.0]

3. Primary Outcome: Percentage of Participants Discontinued From Study Therapy Due to AEs During the DB Treatment Period
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product, was also an AE. For this outcome measure, the primary safety analysis compared the percentage of participants discontinuing study therapy due to an AE in the Immediate Treatment Arm during the double-blinded active treatment period to that of the Deferred Treatment Arm during the double-blinded placebo treatment period.
Time Frame: DB Treatment period (up to Study Week 12)
Population: All randomized participants who received at least one dose of study treatment during the Part A DB period.
Measure: Number; unit: Percentage of Participants
Arm/Group | Immediate Treatment Arm: Grazoprevir/Elbasvir | Deferred Treatment Arm: Placebo > Grazoprevir/Elbasvir
Number analyzed (Participants) | 201 | 100
Percentage of Participants | 0.5 | 1.0
Statistical Analysis 1: Comparison: Immediate Treatment Arm: Grazoprevir/Elbasvir vs Deferred Treatment Arm: Placebo > Grazoprevir/Elbasvir; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Difference in Percentage = -0.5, 95% CI 2-sided [-5.0 to 1.9]

4. Secondary Outcome: Percentage of Participants Achieving Sustained Virologic Response 24 Weeks After the End of All Study Therapy (SVR24)
Description: Blood was drawn from each participant to assess HCV RNA plasma levels using the Roche COBAS® AmpliPrep/COBAS® Taqman HCV Test, v2.0, which has an LLOQ of 15 IU/mL. SVR24 was defined as HCV RNA <LLOQ at 24 weeks after the end of all study therapy. The Clopper-Pearson method was used to construct 95% confidence intervals for the SVR24 rate. The secondary efficacy analysis for Part A evaluated the percentage of participants in the immediate treatment arm (ITA) who achieved SVR24. SVR24 was also calculated for the Deferred Treatment Arm.
Time Frame: 24 weeks after end of all therapy (Study Week 36 for Immediate Treatment Arm and Study Week 52 for Deferred Treatment Arm)
Population: Modified FAS (mFAS): All randomized participants receiving ≥1 dose of active study treatment and excluding participants for study discontinuation for reasons unrelated to treatment regimen, response to HCV treatment, or BL genotype (GT)2, GT3, or GT5. The secondary efficacy analysis was evaluated within participants of the Immediate Treatment Arm.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Immediate Treatment Arm: Grazoprevir/Elbasvir | Deferred Treatment Arm: Placebo > Grazoprevir/Elbasvir
Number analyzed (Participants) | 186 | 85
Percentage of Participants | 94.1 [89.7 to 97.0] | 96.5 [90.0 to 99.3]

ADVERSE EVENTS:
Time Frame: Up to approximately 4 years (Study Week 208)
Description: All-Cause Mortality reported for all randomized participants. AEs reported for all randomized participants receiving ≥1 dose of study treatment. AEs were reported by the treatment that participants were receiving at the time of the event; AEs and deaths for Deferred Group reported separately for placebo (N=100) and active (N=95) treatment periods.
Groups:
- Deferred Treatment Arm: Placebo: In Part A, participants received placebo to MK-5172A once daily for 12 weeks (blinded), followed by 4 weeks of follow-up.
- Deferred Treatment Arm: Grazoprevir/Elbasvir: In Part A, participants received placebo to MK-5172A once daily for 12 weeks (blinded), followed by 4 weeks of follow-up. Afterwards, participants received 12 weeks of open-label treatment with the MK-5172A FDC and were followed-up for 24 weeks. In Part B, participants could enroll in a 3-year follow-up period where they were followed every 6 months for 3 years in an observational cohort (no treatment was administered during Part B).
Arm/Group | Immediate Treatment Arm: Grazoprevir/Elbasvir | Deferred Treatment Arm: Placebo | Deferred Treatment Arm: Grazoprevir/Elbasvir
All-Cause Mortality (participants affected / at risk) | 3/201 | 1/100 | 1/95
Serious Adverse Events (participants affected / at risk) | 16/201 | 4/100 | 7/95
Other Adverse Events (participants affected / at risk) | 108/201 | 46/100 | 36/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Treatment Arm: Grazoprevir/Elbasvir (N=201) | Deferred Treatment Arm: Placebo (N=100) | Deferred Treatment Arm: Grazoprevir/Elbasvir (N=95)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Systemic candida (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Bladder cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ruptured cerebral aneurysm (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Drug abuse (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Hallucination, auditory (Psychiatric disorders) | 1 (3) | 0 (0) | 0 (0)
Personality disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Schizophrenia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Treatment Arm: Grazoprevir/Elbasvir (N=201) | Deferred Treatment Arm: Placebo (N=100) | Deferred Treatment Arm: Grazoprevir/Elbasvir (N=95)
Abdominal pain (Gastrointestinal disorders) | 11 (12) | 4 (4) | 3 (3)
Constipation (Gastrointestinal disorders) | 17 (17) | 4 (5) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 20 (22) | 9 (11) | 8 (8)
Nausea (Gastrointestinal disorders) | 23 (23) | 9 (9) | 8 (8)
Vomiting (Gastrointestinal disorders) | 8 (8) | 7 (7) | 4 (5)
Fatigue (General disorders) | 32 (32) | 20 (22) | 13 (14)
Accidental overdose (Injury, poisoning and procedural complications) | 7 (7) | 4 (5) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8) | 6 (6) | 3 (3)
Headache (Nervous system disorders) | 26 (31) | 14 (20) | 12 (15)
Insomnia (Psychiatric disorders) | 13 (13) | 6 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.